CLINICAL TRIAL: NCT01051609
Title: Prospective Study of Aromatase Inhibitor-Associated Musculoskeletal Symptoms in Non-Metastatic, Post Menopausal Breast Cancer Patients
Brief Title: Aromatase Inhibitor-Associated Musculoskeletal Symptoms in Non-Metastatic, Post Menopausal Breast Cancer Patients
Status: Completed | Type: Observational
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 09-09-058
Record Dates: First submitted 2010-01-15; First posted 2010-01-18 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Breast Cancer
Keywords: Post Menopausal; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Health Records, Personal; Restraint, Physical; Surveys and Questionnaires; Blood Specimen Collection

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Intervention Group: There is only one arm in this trial. Please see interventions for more detailed descriptions.
  Interventions: Other: History and Physical Exam; Other: Grip Strength Measurement; Behavioral: Surveys; Other: Blood Collection; Procedure: Ultrasound of Hand/Wrist

INTERVENTIONS:
Other: History and Physical Exam — The physical exam includes vital signs and ECOG performance status.
Other: Grip Strength Measurement — A hand grip strength test will be used to measure and compare baseline and post-AI treatment forearm muscle strength in each hand.
Behavioral: Surveys — Self-administered surveys including Health Assessment Questionnaire Disability Index, CES-D, FACIT-F, PSQI, GAD7, number of minutes of morning stiffness, and questions pertaining to vasomotor symptoms will be used in this study to assess for presence, severity, characteristics, and associations of AI-associated musculoskeletal symptoms.
Other: Blood Collection — A set of blood markers will be assayed at baseline, 6 months, and 12 months.
Procedure: Ultrasound of Hand/Wrist — An inflammatory arthritis ultrasound scoring method similar to the RAMRIS scoring system used in rheumatoid arthritis, will evaluate joints in the most affected hand and wrist at 6 months.

SUMMARY:
The purpose of this study is to compare pre and post Aromatase Inhibitor (AI) treatment serological markers of inflammation and assess for correlation with AI-MS.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years and older with non-metastatic hormone receptor (ER and/or PR) positive breast cancer who are eligible for and planning on starting treatment with an AI within one month of signing consent.
* Postmenopausal, defined as at least one of the following: a) amenorrhea for at least 12 months b) prior bilateral oophorectomy at least 2 years prior to trial registration.

Exclusion Criteria:

* History of autoimmune connective tissue disease, such as rheumatoid arthritis, lupus, or other autoimmune conditions affecting joints.
* Treatment with steroid (for any condition, except for chemotherapy premedication) within 30 days of trial registration.
* Prior treatment with an AI (patients previously or currently on tamoxifen are eligible as long as patients are off tamoxifen for 2 weeks prior to baseline blood draw)
* Active or ongoing infection
* Known metastatic disease
* Known history of HIV or hepatitis infections
* Ongoing radiation therapy (radiation must have been completed 2 weeks prior to starting treatment with an AI)
* Non-invasive (DCIS, LCIS) cancer only (no diagnosis of invasive cancer)
* Pregnant or lactating
* Unable to speak, read, and write in English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women 18 years and older with non-metastatic hormone receptor (ER and/or PR) positive breast cancer who are eligible for and planning on starting treatment with an AI within one month of signing consent
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2010-05; Primary Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Presence, severity, and change in severity of pain based on joint exam and joint ultrasound inflammatory score. | Study visits at 3, 6, 9 and 12 months after the start of treatment with an Aromatase Inhibitor

CONTACTS AND LOCATIONS:
Overall Officials: Sara Hurvitz, M D, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Jonsson Comprehensive Cancer Center, Los Angeles, California, United States